CLINICAL TRIAL: NCT03304678
Title: Discovery of Sirolimus Sensitive Biomarkers in Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 180003; 18-H-0003
Record Dates: First submitted 2017-10-06; First posted 2017-10-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03-31

CONDITIONS: Lymphangioleiomyomatosis
Keywords: mTORC1 Inhibition; VEGF-D; MicroRNA; Natural History
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with sirolimus (Other): Lymphangioleiomyomatosis (LAM) is a cystic lung disease characterized by proliferation of cells with mutations in the tuberous sclerosis complex (TSC) which leads to activation of the mTORC pathway.
  Interventions: Drug: Sirolimus 2mg

INTERVENTIONS:
Drug: Sirolimus 2mg — Patients with LAM, whose treating physicians have decided that they need to start treatment with sirolimus will be referred to the NIH Clinical Center for these studies.

SUMMARY:
Background:

Lymphangioleiomyomatosis (LAM) is a rare, progressive disease. It usually affects women in the prime of their lives. It typically results in lung destruction. Studies have shown that a drug called sirolimus stabilizes lung function in people with LAM. But researchers do not know what drug dose and blood serum levels are needed to reach this stability. Researchers want to learn more about the right dose of sirolimus for people with LAM.

Objective:

To determine if blood and urine markers after 1 dose and again after 9 months can be used to evaluate the correct dose of sirolimus for people with LAM.

Eligibility:

Women ages 18-90 with LAM whose doctors have decided they should start taking sirolimus to treat it.

Design:

At visit 1, participants will take their first dose of sirolimus by mouth at the clinic. They will have blood and urine collected.

Participants will take 1 tablet of the study drug each day.

Visit 2 will be 3 months after visit 1. Participants will have blood and urine collected.

Visit 3 will be 9 months after visit 1. Participants will have blood and urine collected.

Participant samples will be stored in a secure place. No personal data will be connected to them.

DETAILED DESCRIPTION:
Sirolimus (rapamycin), which acts as a targeted inhibitor of the protein mechanistic target of rapamycin (mTOR), has been shown to be effective in patients with lymphangioleiomyomatosis (LAM). It stabilizes lung function, resolves chylous effusions and lymphangioleiomas and shrinks angiomyolipomas. The current study is to understand better the short-term action of the drug by following the effects on potential biomarkers in blood and urine. Patients with LAM will have samples taken prior to administration of first dose of the drug, at 1 hr and then at 23 hours after the drug (trough level). At 3 and 9 months, samples will be obtained at trough and 1 hour after the dose. Molecular and cellular analyses will be performed to look for potential biomarkers.

ELIGIBILITY:
* INCLUSION CRITERIA
* Female 18 to 90 years of age
* Diagnosis of LAM
* Initiation of sirolimus therapy (2mg daily) based on standard-of-care pulmonary indications and the advice of the patient s local physician

EXCLUSION CRITERIA

* Unable to travel to the NIH
* Unable to provide informed consent
* Advanced stage of a pulmonary or a systemic illness in which the risk of the study is judged to be significant even in the absence of a clear contraindication to the procedures
* Women who are pregnant or lactating

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
to identify if miRNA are responsive to sirolimus in patients with LAM | 9 months
  identify if miRNA are responsive to sirolimus in patients with LAM

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication, whichever comes first, according to Institute policy.
Access Criteria: BioData Catalyst is supported by NHLBI and access to data is controlled by the NHLBI Data Access Committee (DAC) utilizing the database (dbGaP)

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-H-0003.html